CLINICAL TRIAL: NCT01327560
Title: Sleep Quality and Related Factors in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Tso-Hsiao Chen, Department of Nephrology, WanFang Hospital
Other Study IDs: 100003
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Haemodialysis-induced Symptom
Keywords: hemodialysis patients; sleep quality; restless legs syndrome; excessive daytime sleepiness; sleep apnea syndrome
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Restless Legs Syndrome; Disorders of Excessive Somnolence; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sleep quality is an important predictor of healthy status,quality of life and life span. Sleeping problems affect 50%~80% in hemodialysis patients. Sleep quality and related factors research in hemodialysis patients has been discussed and studied globally. Previous studies show insomnia, excessive daytime sleepiness(EDS), sleep apnea syndrome(SAS), restless legs syndrome(RLS) are major causes of poor sleep quality . There is few data to show the influential factors related to sleep quality in Taiwanese hemodialysis patients.

DETAILED DESCRIPTION:
This study will be a cross-sectional design with purposive sample from 2 different dialysis medical centers in Taipei. Two hundred hemodialysis patients meeting inclusion criteria will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient whose age ≧ 20 years old and conscious clear.
* ICD9：585.6
* Every week receives two or three convention hemodialysis treatment above three months.
* May communication with Mandarin or Taiwanese language.
* Patient or caregiver is willing to participate study and sign the inform consent.

Exclusion Criteria:

* Hospitalized hemodialysis patient in recently one month.
* Hemodialysis patient had conscious disturbance, blind or dementia.
* Hemodialysis Patient refuse to interview or fill out questionnaires.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis Patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tso-Hsiao Chen, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan